CLINICAL TRIAL: NCT06963866
Title: A Multicenter, Open-Label, Randomized, Controlled Study of Autologous Stem Cell Transplantation Followed by Anti-BCMA CAR-T Therapy Versus ASCT Alone in Transplant-Eligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Comparing ASCT Followed by Anti-BCMA CAR-T vs. ASCT Alone in NDMM Patients Eligible for ASCT
Acronym: ASCTvsCAR-T
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Chief Hematologist of The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL064-01; XYFY2025-KL064-01 (Other: The Affiliated Hospital of Xuzhou Medical University)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma, Newly Diagnosed
Keywords: Multiple Myeloma; Eligible for ASCT; ASCT; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASCT + CAR-T (Experimental): ASCT followed by BCMA CAR-T
  Interventions: Biological: autologous stem cell transplantation; Biological: CAR-T
- ASCT alone (Active Comparator): ASCT alone, without CAR-T infusion
  Interventions: Biological: autologous stem cell transplantation

INTERVENTIONS:
Biological: autologous stem cell transplantation — Patients in this arm will receive autologous hematopoietic stem cell transplantation (ASCT). Prior to ASCT, the patients underwent 3-4 cycles of induction chemotherapy.
Biological: CAR-T — The T cells are genetically modified to express a chimeric antigen receptor targeting BCMA and are infused 3 days after ASCT at a target dose of ≥2.0×10^6 cells/kg.
  Arms: ASCT + CAR-T

SUMMARY:
This is a prospective study comparing autologous hematopoietic stem cell transplantation followed by anti-BCMA CAR-T to autologous hematopoietic stem cell transplantation alone in the treatment of newly diagnosed multiple myeloma patients.

DETAILED DESCRIPTION:
1. Pre-screening Evaluation. The patient's medical history will be reviewed to assess eligibility based on inclusion criteria. The treatment process and potential risks will be explained, and informed consent will be obtained. Peripheral blood samples will then be collected to test for HIV and to assess the feasibility of CAR-T cell manufacturing. The CAR-T production unit will evaluate the in vitro expansion capacity and transduction efficiency of the patient's T cells within approximately 1-2 weeks to determine whether the patient's peripheral blood is suitable for large-scale CAR-T cell production.
2. Patient Enrollment and Baseline Data Collection. 2.1 Patients who pass the pre-screening will undergo disease assessment and a series of routine evaluations to confirm eligibility for CAR-T cell therapy or autologous hematopoietic stem cell transplantation (ASCT) based on inclusion and exclusion criteria.

   2.2 Required Baseline Tests (within 4 weeks prior to treatment): Complete medical history and physical examination; Electrocardiogram and cardiac function evaluation (MUGA scan or echocardiography); Pulse oximetry to assess lung function; Serum electrolytes and biochemistry; Peripheral blood flow cytometry for quantification of T cells and CD4:CD8 ratio HIV, hepatitis B (HBsAb, HBsAg, HBeAb, HBeAg, HBcAb), and hepatitis C (HCV Ab) screening; Human anti-mouse antibody (HAMA) testing, along with collection of blood and bone marrow samples for DNA extraction and biobanking for future analysis related to tumorigenesis.
3. Autologous Stem Cell Collection and CAR-T Cell Manufacturing. 3.1 Autologous Hematopoietic Stem Cell Collection and Cryopreservation Granulocyte-colony stimulating factor (G-CSF) at 300 μg twice daily for 4 days will be administered. Once peripheral blood CD34+ cells reach the collection threshold, apheresis will be performed with a total blood volume of approximately 6 liters to collect autologous hematopoietic stem cells. The minimum cell dose should be ≥2.0 × 10^6CD34+ cells/kg. DMSO will be added to the collection bag to a final concentration of 20%. The stem cell product will be stored in cryogenic bags, placed in freezing containers, and stored at -80°C.

   3.2 Anti-BCMA CAR-T Cell Manufacturing Apheresis will also be conducted to collect peripheral blood mononuclear cells (PBMCs) for CAR-T cell manufacturing, using approximately 6 liters of blood. Lymphocytes not used for production will be cryopreserved for future research or regulatory review.
4. Conditioning Chemotherapy.

   High-dose melphalan will be used as conditioning therapy beginning 5 days prior to ASCT. The dose ranges from 140-200 mg/m². The purposes of chemotherapy are:

   To reduce tumor burden; To deplete endogenous lymphocytes and facilitate CAR-T cell expansion; To modulate the tumor immune microenvironment. If absolute neutrophil count (ANC) drops below 1.0 × 10^9/L post-chemotherapy, granulocyte colony-stimulating factor (G-CSF) will be administered until ANC exceeds 1.5 × 10^9/L. Antibiotics may be used prophylactically if neutropenia occurs.
5. Post-conditioning Evaluation. Tumor status will be reassessed after conditioning to evaluate baseline disease burden. This includes physical examination, laboratory tests, bone marrow MRD (minimal residual disease) evaluation, and assessment of chemotherapy-related toxicity.
6. Autologous Stem Cell Infusion. Autologous stem cells (minimum 2.0 × 10^6 CD34+ cells/kg) will be reinfused 2 days after conditioning ends. The cryopreserved product will be thawed at 37°C in a water bath and infused intravenously immediately upon full thaw. Vital signs will be closely monitored before, during, and after infusion at 15-minute intervals until the patient stabilizes.
7. Anti-BCMA CAR-T Cell Infusion. CAR-T cells will be infused approximately 3 days after autologous stem cell infusion. The thawed CAR-T product should be infused within 10-15 minutes, with a minimum dose of 2.0 × 10^6 cells/kg. Vital signs will be closely monitored before, during, and after infusion at 15-minute intervals until patient stabilization. Acetaminophen 325-650 mg will be administered orally 30-60 minutes before infusion to reduce infusion-related reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years (inclusive);
2. Estimated life expectancy of more than 12 weeks;
3. Diagnosis of multiple myeloma confirmed by physical examination, pathological evaluation, laboratory tests, and imaging studies;
4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels less than 3 times the upper limit of normal (ULN);
5. Karnofsky Performance Status (KPS) score > 50%.
6. Eligible for ASCT.

Exclusion Criteria:

1. Pregnant or lactating women, or women planning to become pregnant within the next six months;
2. Transduction efficiency of targeted lymphocytes <10%, or expansion fold <5× under CD3/CD28 co-stimulation, as determined by feasibility screening;
3. History of severe allergies or hypersensitivity, especially to interleukin-2 (IL-2);
4. Significant dysfunction of vital organs including the heart, lungs, or brain;
5. Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months after CAR-T infusion
  Progression-Free Survival (PFS) is defined as the time from the date of CAR-T cell infusion to the date of disease progression or death from any cause, whichever occurs first. Disease progression will be determined based on the International Myeloma Working Group (IMWG) criteria. Patients who have not progressed or died will be censored at the date of last follow-up.
Overall Survival (OS) | Up to 36 months after CAR-T infusion
  Overall Survival (OS) is defined as the time from the date of CAR-T cell infusion to death from any cause. Patients who are alive at the time of analysis will be censored at their last known date of follow-up.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months after CAR-T infusion
  Objective Response Rate (ORR) is defined as the proportion of patients achieving a response of partial response (PR) or better, including PR, very good partial response (VGPR), complete response (CR), and stringent complete response (sCR), according to the International Myeloma Working Group (IMWG) criteria. The assessment will be based on laboratory parameters, imaging, and bone marrow evaluation, as applicable.
MRD | Up to 36 months after CAR-T infusion
  The proportion and immunophenotype of plasma cells in bone marrow were analyzed using flow cytometry, with a sensitivity of 10^-5.
Adverse Events (AE) | Up to 36 months after CAR-T infusion
  Focus on adverse events related to ASCT and CAR-T, including CRS, ICANS, coagulation disorders, infections, and other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, Study Chair — The Affiliated Hospital oh Xuzhou Medical University
Locations (1):
- The Affiliated Hospital oh Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No